CLINICAL TRIAL: NCT00680667
Title: Phase I Clinical Trial of Trametes Versicolor in Women With Breast Cancer
Brief Title: Clinical Trial of Trametes Versicolor in Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007LS019; U19AT001998 (NIH); UMN-0611M96168 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2008-05-18; First posted 2008-05-20 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — VPS Coriolus versicolor extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trametes Versicolor (Experimental): Females with Stage I-III infiltrating ductal adenocarcinoma of the breast being treated with Trametes versicolor capsules for 6 weeks after receiving radiation therapy.
  Interventions: Biological: Coriolus versicolor extract

INTERVENTIONS:
Biological: Coriolus versicolor extract — Trametes versicolor (Tv) capsules at the assigned dose level (3 grams/day up to 24 grams/day) twice a day every day and continuing for weeks.
  Other Names: T. versicolor; Tv; turkey tail

SUMMARY:
RATIONALE: Coriolus versicolor mushroom extract may slow the growth of cancer cells and may be an effective treatment for breast cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of coriolus versicolor extract in treating women with stage I, stage II, or stage III breast cancer who have finished radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of oral coriolus versicolor extract in women with stage I-III, estrogen receptor- and/or progesterone receptor-negative or positive (as of 1/26/2009), infiltrating ductal adenocarcinoma of the breast who have recently completed standard post-surgery radiotherapy.

Secondary

* To determine the feasibility of measuring changes in fatigue and quality of life of patients treated with this drug.
* To characterize the toxicity of this drug in these patients.
* To gather preliminary data that compare baseline and post-treatment immunologic measures, including differential blood counts (i.e., WBC), natural killer cell activity, phagocytic index, regulatory cell assay, T/B/NK cell population subset assays, peripheral blood mononuclear cell production of levels of interferon gamma, and tumor necrosis factor-alpha in these patients.

OUTLINE: Patients receive oral coriolus versicolor extract twice daily for 6 weeks.

Patients undergo quality of life and fatigue assessment at baseline, weekly during study, and at the 3-week follow-up visit.

Blood samples are collected periodically for immunological marker studies. Samples are analyzed for T-regulatory cell, T-and B-lymphocyte, and NK cell activity in peripheral blood mononuclear cells (PBMC), phagocytic index in monocytes and granulocytes, and cytokine secretion and upregulation by flow cytometry, cytotoxicity assays, cytolysis assays, T-regulatory cell assay, or T/B/NK cell population subset assays. Changes in the production of tumor necrosis factor-alpha and interferon-gamma in serum and in supernatants of PBMCs are analyzed via standard enzyme-linked immunosorbent assay.

After completion of study treatment, patients are followed at 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis, within the previous 12 months with Stage I-III, infiltrating ductal adenocarcinoma of the breast who have undergone surgery and chemotherapy and are able to begin study treatment within 5 days after the last dose of radiotherapy
* Estrogen and/or progesterone receptor-negative or positive
* Willing to eat consistent diet throughout the study, and avoid dietary sources of mushrooms
* Willing to avoid taking any product containing Trametes versicolor, other immune modulating medicinal mushrooms, or other herbal products believed to have immune modulating effects, during radiotherapy and until completion of the subject's last clinic visit on the study.
* Adequate organ function within 14 days of study enrollment including the following:

  * Adequate bone marrow reserve: White blood cells (WBC) ≥ 2,000/mm³, Platelet count ≥ 100,000/mm³, Hemoglobin ≥ 9 g/dL
  * Hepatic: Bilirubin ≤ 20% times upper limit of normal (ULN), Alkaline phosphatase ≤ 20% times ULN, AST and ALT ≤ 20% times ULN
  * Renal: Creatinine ≤ 20% times ULN
  * Nutritional status: Albumin ≥ 3.0 g/dL
* Negative pregnancy test
* Voluntary written consent before performance of any study-related procedure not part of the normal medical care

Exclusion Criteria:

* Pregnant - Patients with reproductive potential must use an approved non-hormonal contraceptive method if appropriate during and for 4 weeks after the last dose of Trametes versicolor.
* Known allergy to fungi, including mushrooms
* Serious concurrent medical or psychiatric disorder (e.g., active infection or uncontrolled diabetes) that, in the opinion of the investigator, would compromise the safety of the patient or the patient's ability to complete the study
* Receipt of hematopoietic growth factors (e.g., Neupogen™, Epogen™) within the previous 4 weeks
* Unwilling to maintain consistency in type and dose of concurrent complementary and alternative medicine therapies
* Unwilling to discontinue excluded medications and supplements

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 6 Weeks After Treatment

SECONDARY OUTCOMES:
Quality of life | Over 6 Weeks
  as measured by the Functional Assessment of Cancer Therapy-for Patients With Breast, v4.0, questionnaire. The FACT-B is a 37-item quesionnaire using a 5-point Likert scale that evaluates physical well-being, social/family well-being, emotional well-being, functional well-being and additional concerns of breast cancer patients.
Fatigue | Over 6 Weeks
  as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue, v4.0, questionnaire. The FACIT-Fatigue is a 13 item fatigue scale collected at baseline, weekly and 6 weeks, and at the 3 week follow-up visit.
Symptom Assessment | Weekly and at 3 Week Follow-Up
  Toxicity will be assessed by the NCI CTCAE v3.0 (see Adverse Event section). The Symptom Assessment questionnaire is completed weekly during study and once at the 3-week follow-up visit
NK cell activity | Over 6 weeks
  Percent change in NK cell activity associated with coriolus versicolor extract
comparison of immunologic measures | Baseline and Post-Treatment
  Will be performed by collecting peripheral blood at baseline, weeks 2,4,6 and 9 during study.
  Preliminary data that compare baseline and post-treatment immunologic measures including natural killer cell activity, phagocytic index, T regulatory cell assay, T/B/NK cell population subset assays, and cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Torkelson, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Bastyr University, Kenmore, Washington